CLINICAL TRIAL: NCT06323187
Title: Optimization of Cervical Collections in Pregnancy
Acronym: OCCP
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Sascha Drewlo (Other)
Responsible Party: Sponsor-Investigator, Dr. Sascha Drewlo, Professor, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 4656
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cervix; Pregnancy; Inherited Genetic Conditions (Diagnosis); Preeclampsia; Fetal Growth Retardation
MeSH Terms: conditions — Disease; Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Cervical specimens collected from the uterine cervical canal, similar to collection for a PAP test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Participants: Pregnant participants will be randomly assigned to provide a cervical sample using one of the devices/procedures for cervical fluid collection.
  Interventions: Diagnostic Test: Cervical Sampling
- Non-Pregnant Participants: Non-pregnant participants will be randomly assigned to provide a cervical sample using one of the devices/procedures for cervical fluid collection.
  Interventions: Diagnostic Test: Cervical Sampling

INTERVENTIONS:
Diagnostic Test: Cervical Sampling — Each participant will provide a sample of fluid or mucus collected from the uterine endocervix.

SUMMARY:
Fetal cells are not easily obtained from pregnant patients; this curtails testing to assess the health of the fetus and the mother. Currently, the only way of diagnosing fetal genetic or chromosomal abnormalities is by invasive techniques, such as chorionic villous sampling (CVS) and amniocentesis performed at 10 to 13 weeks and after 15 weeks of gestation, respectively. Although small, there is a risk for fetal loss with these procedures. Transcervical cell sampling (TCS), similar to a Pap smear, is a platform that meets the requirements for prenatal genetic testing (genetic testing with fetal cells obtained before birth), as well as diagnosis of maternal pregnancy complication, at a very early stage of pregnancy (as early as 5 weeks) and carries low risk for the mother and the developing fetus.

This study will examine cervical fluid collected using various noninvasive methods for TCS in pregnant women. The number of placental cells will be assessed against similarly obtained samples from nonpregnant women of reproductive age who lack cells derived from a placenta. Participating volunteers will provide written informed consent. Only standard medical procedures and approved devices will be used for collection of cervical fluid, minimizing risk to the participants and their fetuses. No test results or other benefits will be available to the participants.

DETAILED DESCRIPTION:
The study will be non-interventional and designed for prospective sample collection and concurrent analysis. The primary endpoint will be a determination of the number of extravillous trophoblast (EVT) cells (placental cells that migrate into the reproductive tract) obtained by each device and procedure. The number of EVT cells, adjusted for purity (expression of a fetal marker, e.g., cytokeratin 7) directly determines the amount of fetal DNA that will be available for prenatal genetic testing. Secondary endpoints will include the total number of cells in the initial cervical samples and the amount of fetal DNA, RNA and/or protein isolated from the EVT cells. Where fetal DNA is obtained, we will sequence the fetal and maternal DNA for comparison of single nucleotide variant (SNV) and short tandem repeat (STR) loci to assess the purity of the fetal DNA (fetal fraction) or perform whole genome sequencing. Cell-free biomolecules present in cervical fluid will also be assessed for proteins or RNAs associated with adverse pregnancy outcomes, or cell-free fetal DNA. These parameters will be compared between the various collection methods to describe an optimal collection protocol for the purpose of analyzing fetal cells and their components.

Cohort: We will follow a group of pregnant individuals over time, collecting cervical secretions at various stages throughout pregnancy and then comparing these data to the pregnancy outcomes.

Control: We will collect cervical fluid from non-pregnant, non-menstruating women of reproductive age for comparison to the cohort participant samples. It is expected that cells or biomolecules produced by the placenta will be absent and that any signals detected would define background levels.

Descriptive: The study aims to observe and describe the properties of cervical secretions throughout pregnancy and their association with pregnancy outcomes or fetal genotype.

Establishing a registry/database: The researchers need to create a database to organize and analyze the information collected from participants, such as the properties of their cervical secretions and the outcomes of their pregnancies.

Pregnant women (N=2000) will be enrolled in this study because it is an investigation of a method for prenatal testing and the endpoint is detection of EVT cells or their products that are of fetal origin, specifically from the placenta. The age range of 18 to 45 years was chosen because this is the principal range for reproductive activity in women. Nonpregnant women (N=600) will also be enrolled to control for EVT cells in pregnant samples and determine the respective number of cells obtained in the study protocol when no EVT cells are present.

There will be no enrollment restriction based on racial or ethnic origins. The aim is to include sufficient diversity in enrollment to ensure that the benefits and burdens of research participation are distributed in an equitable manner. It is also desirable that the findings are reproducible across all racial and ethnic groups.

If the sample is taken at the time of a Pap smear, the healthcare professional will follow recommended procedures. The initial excess mucus from the canal and ectocervix, will be deposited in the collection containers provided by the PI rather than being discarded. If sample collection is conducted at a different time than the pregnancy cervical cytology, a cervical brush in addition may be obtained. Sample collection kits using devices used for Pap smears (including during pregnancy) and other methods to be investigated will be provided to the clinics. These kits will contain all devices for sample collection and shipment back to the PI. Kits will also contain a participant data sheet and instructions for sample collection. All kit materials will be coded to identify each participant. The key to the codes will be retained by each clinical site collaborator in a locked cabinet in their office so that personnel working with the PI will only have the de-identified code for each participant. To link laboratory data to clinical data, the clinical site collaborator will conduct the analysis using the key to the codes. No information from the analysis of the cervical fluid will be returned to the participant or their doctor since the study is designed to evaluate the procedures for sample procurement, not the test results.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy Before 30w0d gestation for pregnant participants
* Regular menses within previous month for non-pregnant participants
* 18-45 years old

Exclusion Criteria:

* Bleeding >5 days in first trimester for pregnant participants
* Ruptured membranes for pregnant participants
* Currently menstruating for non-pregnant participants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women age, 18-45 who are either pregnant before 30w0d gestation or non-pregnant and not menstruating.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Cellular content | 2 weeks
  The number of cells in the cervical sample that express markers for extracellular trophoblast will be determined.
Cell-free content | 2 weeks
  The concentration of placental biomarkers (e.g., HLA-G, KRT7) in the cell-free supernatant of the cervical sample will be determined. Also nucleic acids derived from the placenta, including fetal DNA and placental RNAs.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Drewlo, PhD, Principal Investigator — Sunnybrook Research Institute

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD outside of the study team as per institutional REB guidelines. Any researchers wishing to access study IPD can contact the PI.

REFERENCES:
- [Background] Practice Bulletin No. 162: Prenatal Diagnostic Testing for Genetic Disorders. Obstet Gynecol. 2016 May;127(5):e108-e122. doi: 10.1097/AOG.0000000000001405. PMID 26938573
- [Background] Drewlo S, Armant DR. Quo vadis, trophoblast? Exploring the new ways of an old cell lineage. Placenta. 2017 Dec;60 Suppl 1(Suppl 1):S27-S31. doi: 10.1016/j.placenta.2017.04.021. Epub 2017 Apr 26. PMID 28483162
- [Background] Moser G, Drewlo S, Huppertz B, Armant DR. Trophoblast retrieval and isolation from the cervix: origins of cervical trophoblasts and their potential value for risk assessment of ongoing pregnancies. Hum Reprod Update. 2018 Jul 1;24(4):484-496. doi: 10.1093/humupd/dmy008. PMID 29608700